CLINICAL TRIAL: NCT05384080
Title: Prospective, Non-interventional, Observational Study in Patients With IBD Receiving IV or SC Vedolizumab Therapy to Observe Route of Administration Choices and Outcomes (VARIETY-POLAND)
Brief Title: A Study in Adults With Ulcerative Colitis (UC) or Crohn's Disease (CD) Receiving Vedolizumab in Real-World Practice in Poland
Acronym: VARIETY
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: VedolizumabSC-4004
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Disease (IBD); Crohn's Disease; Ulcerative Colitis
Keywords: Drug Therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With IBD: Participants diagnosed with moderately to severely active IBD (UC or CD) who are currently ongoing vedolizumab IV induction treatment in accordance with the current Summary of Product Characteristics (SmPC) and National Drug Program (NDP) at baseline or receiving vedolizumab ongoing or maintenance IV treatment with the option to switch to vedolizumab SC treatment, will be observed prospectively for 24 months.

SUMMARY:
The primary reason of this study is to observe current treatment options in participants receiving Vedolizumab, intravenous (IV) or subcutaneous (SC), for IBD in Poland. There is no treatment involved in this study, this is only an observational review of ongoing/initiating treatment data relating to Vedolizumab induction and maintenance treatment for IBD [including Ulcerative Colitis (UC) and Crohn's Disease (CD)].

DETAILED DESCRIPTION:
This is a non-interventional, prospective study of participants with moderately to severely active IBD (UC or CD) who are initiating or currently ongoing induction or maintenance treatment with vedolizumab in the real world setting.

The study will enroll approximately 160 participants: 100 participants with UC and 60 participants with CD. The data will be collected prospectively at the study sites and will be recorded into electronic case report forms (e-CRFs). All the participants will be assigned to a single observational cohort:

•Participants with IBD

This single center study will be conducted in Poland at public hospitals and institutions that treat UC and CD. The overall duration of the study will be at least 24 months. Data will be collected at baseline, every 3 months within the first year and every 6 months within the second year, and at the time of switch, discontinuation and/or at routine follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1.Participants with moderately to severely active IBD (UC or CD), initiating or ongoing IV induction treatment with vedolizumab in accordance with the current SmPC and National Drug Program (NDP) at baseline OR IBD participants receiving ongoing/maintenance IV vedolizumab treatment, with the option to switch to SC vedolizumab maintenance treatment.

Exclusion Criteria:

1. Prior history of intolerability, hypersensitivity, or other contraindications (active severe infections such as tuberculosis, sepsis, cytomegalovirus, listeriosis, and opportunistic infections such as Progressive Multifocal Leukoencephalopathy) to vedolizumab therapy as defined in the current SmPC.
2. Current or planned participation in an interventional clinical trial for CD or UC.
3. Cognitive incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

   .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with moderately to severely active UC or CD receiving vedolizumab treatment in accordance with the approved SmPC and NDP.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Persisting on Treatment With Vedolizumab IV Compared to Participants With Treatment Change up to 24 Months | Baseline up to 24 months
Time to any Treatment Change | Baseline up to 24 months
Number of Participants Who Discontinued Vedolizumab Treatment | Baseline up to 24 months
Number of Participants With Reason for Treatment Change | Baseline up to 24 months
Number of Participants With Change in Vedolizumab Dosing Frequency | Baseline up to 24 months
Number of Participants Who Changed to Another Treatment | Baseline up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- Poland (11):
  - Uniwersytecki Szpital Kliniczny, Wroclaw, Dolnoslskie
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej W Miedzychodzie, Międzychód, Greater Poland Voivodeship
  - Szpital Kliniczny Im. Heliodora Swiecickiego Uniwersytetu Medycznego Im. Karola Marcinkowskiego W Poznaniu, Poznan, Greater Poland Voivodeship
  - Szpital Uniwersytecki Nr 2 Im. Dr Jana Biziela W Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Szpital Uniwersytecki w Krakowie, Krakow, Lesser Poland Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 W Lublinie, Lublin, Lublin Voivodeship
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw, Masovian Voivodeship
  - Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie, Warsaw, Masovian Voivodeship
  - Wojskowy Instytut Medyczny, Warsaw, Masovian Voivodeship
  - HT Centrum Medyczne, Tychy, Slskie
  - Spzoz Uniwersytecki Szpital Kliniczny Nr 1 Im. Norberta Barlickiego Uniwersytetu Medycznego, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click on this link. — https://clinicaltrials.takeda.com/study-detail/8b74558af8a3453a?idFilter=%5B%22VedolizumabSC-4004%22%5D